CLINICAL TRIAL: NCT07264140
Title: Assessing and Improving Misuse of Inhalers in Outpatients With COPD - The AIMO COPD Study
Brief Title: Assessing and Improving Misuse of Inhalers in COPD Outpatients
Acronym: AIMO COPD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital Fribourgeois (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AIMO-COPD
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; Chronic Obstructive Pulmonary Disease; Inhaler Technique; Inhaler Misuse; Peak Inspiratory Flow; Inhaler Education; Inhaler Optimization; Respiratory Physiotherapy; In-Check DIAL; Outpatient COPD Care
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned in a 1:1 ratio to either a structured, physiotherapist-led inhaler-optimization program or to usual outpatient COPD care. Both groups complete identical baseline and 12-month assessments, but only the intervention group receives three physiotherapist visits focused on inhaler technique review, peak inspiratory flow measurement, and individualized teach-to-goal education. Outcome assessors at Month 12 are blinded to group allocation.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants receive a structured, physiotherapist-led inhaler-optimization program in addition to their usual COPD care. The program includes three in-person visits at approximately Months 3, 6, and 9. During each visit, the physiotherapist assesses inhaler technique using device-specific placebo inhalers, measures peak inspiratory flow (PIF) with the In-Check DIAL® device, and provides individualized teach-to-goal inhaler education. If persistent critical errors or suboptimal PIF are identified, a recommendation is made to the treating physician to adapt the inhaler type. All participants undergo baseline and 12-month assessments identical to the control group.
  Interventions: Behavioral: Physiotherapist-Led Inhaler Optimization Program
- Usual Outpatient COPD Care (No Intervention): Participants receive standard outpatient COPD management from their treating physician. Usual care may include medication adjustments and inhaler review at the physician's discretion, but no structured physiotherapy sessions are added. Participants complete baseline and 12-month assessments identical to the intervention group, including inhaler technique evaluation, PIF measurement, respiratory questionnaires, and lung function testing.

INTERVENTIONS:
Behavioral: Physiotherapist-Led Inhaler Optimization Program — This intervention consists of a structured, physiotherapist-led inhaler-optimization program delivered over 12 months in addition to usual outpatient COPD care. Participants attend three face-to-face sessions at approximately Months 3, 6, and 9. During each session, a trained physiotherapist evaluates inhaler technique using device-specific placebo inhalers and validated checklists, measures peak inspiratory flow (PIF) with the In-Check DIAL® device adjusted to the resistance of each inhaler, and provides individualized teach-to-goal education with iterative demonstration and feedback until correct technique is achieved. If the participant continues to demonstrate critical errors or cannot generate an adequate PIF for their prescribed device, the physiotherapist notifies the treating physician and recommends adapting the inhaler type. The intervention does not include medication changes or pharmacologic treatment; it focuses specifically on optimizing device handling and matching inhal
  Arms: Intervention Group

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a common long-term lung disease that causes breathlessness, cough, and frequent flare-ups. Most patients with COPD use inhaled medications every day. However, many people do not use their inhalers correctly, or they cannot generate the right inspiratory flow for their device. When inhalers are used incorrectly, the medication does not reach the lungs properly, symptoms worsen, and the risk of exacerbations increases.

The goal of this study is to determine whether a structured inhaler-optimization program can reduce incorrect inhaler use in outpatients with COPD. The program is delivered by trained physiotherapists over 12 months and includes three in-person sessions. During these sessions, the physiotherapist evaluates the patient's inhaler technique using placebo devices, measures the patient's peak inspiratory flow with the In-Check DIAL® device, and provides individualized "teach-to-goal" education to help patients use their inhalers correctly. If the patient continues to make critical errors or cannot generate the appropriate inspiratory flow for their inhaler, the physiotherapist may recommend adapting the type of inhaler to better match the patient's abilities.

Participants will be randomly assigned to one of two groups. The intervention group will receive the structured program in addition to their usual COPD care. The control group will continue with usual outpatient care without the physiotherapist-led sessions. All participants will complete baseline and 12-month assessments, which include inhaler technique evaluation, inspiratory flow measurement, respiratory questionnaires, and lung function tests. Telephone follow-up calls will be performed at months 2, 5, and 8 to monitor symptoms, inhaler use, and adherence.

The main outcome of the study is the proportion of inhalers used incorrectly at 12 months. Incorrect use is defined as at least one critical inhaler technique error or an inspiratory flow that is too low or too high for the patient's device. Secondary outcomes include changes in respiratory symptoms, health status, adherence to inhaled treatment, patient satisfaction with inhalers, confidence in inhaler use, and the number of COPD exacerbations or hospitalizations during the study.

This research may help improve everyday inhaler use in people with COPD and support more personalized inhaler selection in routine clinical care. Although participants may not benefit directly, the study poses minimal risks and may contribute to future improvements in COPD management.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a major cause of morbidity and mortality worldwide. Most patients rely on inhaled medications to control symptoms and reduce the risk of exacerbations. However, many patients do not use their inhalers correctly. Critical errors-such as incorrect preparation of the device, improper inhalation technique, or an inspiratory flow that is not appropriate for the device-are common and can lead to reduced drug delivery, poorer symptom control, and more frequent exacerbations. Previous studies conducted at the study site have shown that nearly 70% of hospitalized COPD patients used at least one inhaler incorrectly. In addition, peak inspiratory flow (PIF) varies between individuals, and many patients are unable to generate the flow required for certain dry powder inhalers. Despite this, regular assessment of inhaler technique and inspiratory flow is not systematically implemented in outpatient practice.

This randomized controlled trial evaluates whether a structured, physiotherapist-led inhaler-optimization program can reduce incorrect inhaler use among outpatients with COPD. The intervention includes three face-to-face visits over 12 months. During these sessions, physiotherapists trained in inhaler technique assessment use device-specific placebo inhalers and standardized checklists to identify critical errors. They also measure PIF with the In-Check DIAL® device, adjusted to the resistance of each patient's inhaler. The physiotherapist then provides individualized "teach-to-goal" education, with demonstration, correction, and repeated practice until mastery of the inhaler technique is achieved. When persistent errors or suboptimal PIF are identified, the physiotherapist informs the treating physician to consider adapting the type of inhaler.

Participants are randomly assigned (1:1) to the intervention group or the usual-care group. Usual care consists of regular management by the treating physician, which may include inhaler review at the physician's discretion, but without the structured physiotherapist-led sessions. Both groups undergo baseline and 12-month assessments that include inhaler technique evaluation using placebo devices, PIF measurement, respiratory questionnaires, and pulmonary function testing. Participants in both groups also receive telephone follow-up calls at months 2, 5, and 8 to assess symptoms, inhaler use, adherence, and confidence in inhaler use.

The primary endpoint is the proportion of misused inhalers at 12 months. An inhaler is considered misused if the patient demonstrates at least one critical technique error or if their measured PIF is outside the recommended range for their specific device. This composite outcome captures both aspects of inhaler adequacy: correct handling of the device and physiological ability to use it effectively. Secondary endpoints include changes in health status measured by validated respiratory questionnaires (CAT and CCQ), treatment adherence using the TAI questionnaire, satisfaction with inhalers, confidence in inhaler use, pulmonary function parameters, and the number of COPD exacerbations and hospitalizations over the 12-month follow-up.

The trial uses a pragmatic design to reflect real-world outpatient care. The inhaler-optimization program is intended to be simple, scalable, and easily integrated into routine COPD management. The educational approach is based on individualized instruction and repeated reinforcement, which patients in prior studies have reported as highly valuable. Outcome assessment at 12 months is performed by assessors who are not involved in delivering the intervention and are instructed to remain blinded to group allocation.

The study is minimal-risk and non-invasive. Potential risks include temporary fatigue or coughing during repeated inspiratory maneuvers and the time required for study visits and follow-up calls. The intervention does not involve investigational products or exposure to radiation. Data are collected according to Swiss data protection regulations using coded identifiers and secure REDCap databases.

By evaluating inhaler technique and inspiratory flow in a structured, standardized manner, this study aims to provide new evidence on how to improve inhaler use in COPD. Results may support more personalized device selection, enhance patient education practices, and reduce COPD exacerbations and associated healthcare burden. The findings may be applicable to a wide range of outpatient settings and could inform future guidelines on inhaler optimization in chronic respiratory diseases.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 years or older
* Confirmed diagnosis of COPD by spirometry (FEV₁/FVC < 0.7)
* Current use of at least one maintenance inhaler
* Follow-up in the outpatient pneumology clinic of HFR Fribourg
* Ability to provide written informed consent

Exclusion Criteria:

* Inability to provide informed consent (e.g., severe cognitive impairment, advanced psychiatric disorder, unresolved language barrier)
* Life expectancy of less than 12 months
* Presence of another predominant chronic lung disease (e.g., asthma, interstitial lung disease, pulmonary fibrosis)
* Contraindication to participation (e.g., severe motor impairment preventing inhaler handling)
* Participation in another interventional trial related to inhaler technique

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2026-03-02 (Estimated); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of Misused Inhalers at 12 Months | Month 12
  An inhaler is classified as misused if the participant demonstrates at least one critical inhaler technique error or if the measured peak inspiratory flow (PIF) is outside the recommended range for the specific device. Critical errors are assessed using device-specific standardized checklists with placebo inhalers. PIF is measured using the In-Check DIAL® device set to the resistance of each inhaler. The first PIF measurement, reflecting the participant's usual inhalation technique, is used to classify misuse. Device-specific thresholds define insufficient PIF for dry powder inhalers and excessive PIF for pMDIs or soft-mist inhalers.

SECONDARY OUTCOMES:
Change in COPD Assessment Test (CAT) Score | Baseline and 12 months
  Change in health status measured with the COPD Assessment Test (CAT), a validated 8-item questionnaire (score range 0-40, higher scores indicate worse symptoms). The change from baseline to Month 12 will be compared between groups.
Change in Adherence to Inhaled Therapy (TAI Score) | Baseline and 12 months
  Change in adherence measured with the Test of Adherence to Inhalers (TAI), a validated tool assessing intentional and unintentional non-adherence. Total score 10-50, higher scores indicate better adherence.
Change in Patient Satisfaction With Inhalers (FSI-10 Score) | Baseline and 12 month
  Satisfaction with inhaler devices assessed using the 10-item Feeling of Satisfaction with Inhaler (FSI-10) questionnaire. Higher scores indicate greater satisfaction.
Change in Confidence in Inhaler Use | Baseline and 12 months
  Change in confidence using a 7-point Likert-type scale ranging from 0 (no confidence) to 7 (complete confidence). Measured at baseline and Month 12 to assess improvement in inhaler self-efficacy.
Change in Pulmonary Function Parameters | Baseline and 12 months
  Change in post-bronchodilator FEV₁ (liters and % predicted), FEV₁/FVC ratio, and FEF25-75%, measured according to ATS/ERS standards. Comparison of changes from baseline to Month 12 between groups.
Time to First COPD Exacerbation | Up to 12 months
  Time from randomization to the first COPD exacerbation requiring systemic corticosteroids, with or without antibiotics. Exacerbations are confirmed through medical records or treating physician.
Time to First COPD-Related Hospitalization | Up to 12 months
  Time from randomization to the first unplanned hospital admission for a COPD exacerbation, confirmed through discharge documentation.

CONTACTS AND LOCATIONS:
Locations (1):
- HFR Fribourg, Fribourg, Switzerland

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. The study involves coded health-related data collected at a single center, and the protocol does not include provisions for external data sharing. Data are stored securely on HFR servers according to Swiss data protection regulations (HRA and FADP) and are retained only for the purposes of the approved study. Any future secondary use would require additional ethics approval and, if applicable, new participant consent.